CLINICAL TRIAL: NCT06383143
Title: Promoting Diagnosis and Management of AL in Italy (ProDigALIty)
Acronym: ProDigALIty
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giovanni Palladini, MD, PhD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: AC-020-IT
Record Dates: First submitted 2024-04-19; First posted 2024-04-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-07

CONDITIONS: AL Amyloidosis; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with MGUS and aFLCR and with SMM: Part A: Patients with MGUS and aFLCR and patients with SMM undergoing an active, biomarker-based screening of presymptomatic amyloid organ involvement.
  Part B: Newly diagnosed patients with AL amyloidosis identified through Part A or with clinically overt AL amyloidosis evaluated in the frame of routine clinical assessments and referred to the Amyloidosis Research and Treatment Center in Pavia or managed locally at the participating Italian Hematologic Departments
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The investigators plan to establish a dedicated network of Italian Hematologic Departments interconnected with the Amyloidosis Research and Treatment Center in Pavia to:

1. Implement a biomarker-based screening strategy to promote early diagnosis of AL amyloidosis among at-risk patients, including patients with monoclonal gammopathy of undetermined significance, MGUS, and altered free light chain ratio (aFLCR), and patients with smoldering multiple myeloma (SMM)
2. Expedite and facilitate patients' referral and their enrollment in ongoing pre-clinical/clinical studies, also to reflect a broader spectrum of the real-world population of patients with AL amyloidosis in Italy;
3. Investigate the clinical utility of novel diagnostic technologies, including light chain sequencing and N-glycosylation analysis

DETAILED DESCRIPTION:
AL amyloidosis (AL) is a rare, severe protein conformational disease caused by misfolding and extracellular deposition of patients-specific monoclonal immunoglobulin light chains in form of amyloid fibrils. This process can affect virtually any body site and result in potentially fatal organ dysfunction.

In a significant proportion of cases, AL is diagnosed late, when advanced, often irreversible organ involvement limits therapeutic options and greatly limits survival. Thus, efforts at promoting early diagnosis are urgently needed.

The presence of a monoclonal protein (M protein) or an abnormally increased concentration of serum free LCs (FLCs) invariably precedes clinically overt AL amyloidosis by several years. Moreover, about 95% of patients with AL have an altered FLC ratio (FLCR) at diagnosis. Yet, AL is often diagnosed late also in patients with known monoclonal gammopathy under hematological follow-up. Screening of at-risk patients with biomarkers of early amyloid organ involvement has been advocated, but not largely implemented.

Diagnosis and management of AL patients require access to sophisticated technologies and expertise available at large tertiary Amyloid Centers. Yet, new models of patients' care are required to intercept those patients who cannot travel to distant, tertiary centers, in order to provide state-of-the-art care to all and to be able to analyze and describe the natural history of the disease in a contemporary, real-world setting.

New molecular features associated with the propensity of light chains to form amyloid are emerging, but their potential clinical utility is unknown. Building on >30 years-experience of the Italian Referral Center for Systemic Amyloidoses and leveraging on an already existing disease registry and a one-of-a-kind biorepository of clinically annotated biological samples, the study plans to extend and corroborate the activity of the Italian Amyloidosis Network, through the involvement of large Hematology Departments strategically distributed across the Country and the establishment of a structured program of patients' referral and sample/data transfer.

The study will be conducted as follows:

Part A: an active biomarker-based surveillance of pre-symptomatic signs of amyloid organ involvement in at-risk subjects (patients with MGUS and aFLCR and patients with SMM) will be implemented in the participating Italian Hematologic Departments. This will enable the verification of the feasibility of such biomarker-based screening, allow the description of baseline characteristics of at-risk patients, and promote early diagnosis of AL amyloidosis.

Part B: newly diagnosed AL amyloidosis patients (either from Part A or from patients with clinically overt AL amyloidosis evaluated in the frame of routine clinical assessments) will be either referred to the Amyloidosis Research and Treatment Center in Pavia or managed locally, with clinical data prospectively entering a disease registry and diagnostic leftovers from biospecimens stored in a biorepository. This will aim to increase referral and increment inclusion of real-world cases of AL amyloidosis in the disease registry and linked biorepositories, as well as patients' enrollment in other already approved and funded pre-clinical and clinical studies on basic disease mechanisms, as well as new diagnostic/therapeutic approaches in AL amyloidosis.

Part C: exploiting data collected from patients enrolled in both part A and part B, the clinical utility of clonal light chain profiling (including light chain sequencing, evaluation of the N-glycosylation status, and artificial intelligence-based amyloidogenicity prediction) will be assessed.

ELIGIBILITY:
PART A

Inclusion Criteria:

* diagnosis of MGUS with altered FLCR or SMM;
* treatment-naïve;
* age ≥18 years;
* ability to understand and willingness to sign an informed consent;
* planned follow-up at participating center.

Exclusion Criteria:

* Diagnosis of symptomatic monoclonal gammopathies;
* Previous treatment for monoclonal gammopathies.

PART B

Inclusion criteria:

* diagnosis of systemic AL amyloidosis;
* treatment-naïve;
* age ≥18 years;
* ability to understand and willingness to sign an informed consent;
* planned follow-up at participating center.

Exclusion criteria:

* non-AL amyloidosis;
* previous treatment for AL amyloidosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participating Departments of Hematology will be involved in screening at-risk patients with monoclonal gammopathies and refer suspected/confirmed AL cases to the Amyloidosis Center in Pavia.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Assess proportion of patients with newly diagnosed AL identified through the biomarker-based screening of at-risk patient | 2 years
  Part A of the study: the proportion of patients with newly diagnosed AL through the biomarker-based screening of at-risk patients with a known monoclonal gammopathy will be identified.
Assess the proportion of patients with deep haematological response after frontline therapy (best response evaluation) in the new enhanced, contemporary, real-world series of AL patients enrolled during the study. | 2 years
  Part B of the study: The proportion of patients with deep hematological response after frontline therapy will be assessed
3. Identify associations of clonal light chain features with different clinical features at baseline. | 2 years
  Part C of the study: Associations of clonal light chain features with different clinical features at baseline, including organ tropism and clonal burden, will be assessed.

SECONDARY OUTCOMES:
Description of the baseline characteristics and 6-months outcome, as well as the time to AL development for patients with AL identified through the biomarker-based screening | 6 months
  Part A: the baseline characteristics and 6-months outcome, as well as the time to AL development for patients with AL identified through the biomarker-based screening will be evaluated
Description of the baseline characteristics of MGUS/SMM patients with abnormal FLCR | 2 years
  Part A: the baseline characteristics of MGUS/SMM patients with abnormal FLCR will be described
Identification of clinical and biological correlates of hematological response | 2 years
  part B: clinical and biological correlates of hematological response will be identified
To verify whether implementing a dedicated pipeline for referral of AL patients to the National Referral Center will increase the proportion of patients from spoke centers | 2 years
  Part B: it will be verified if implementing a dedicated pipeline for referral of AL patients to the National Referral Center will increase the proportion of patients from spoke centers
Identification of associations of clonal light chain features with event-free survival | 2 years
  Part C: associations of clonal light chain features with event-free survival will be identified.
Validation of existing algorithms for predicting AL amyloidosis status | 2 years
  Part C: The diagnostic performance of existing algorithms for predicting clonal light chain amyloidogenicity will be evaluated.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Policlinico Consorziale, Bari
  - Azienda Ospedaliero Universitaria Policlinico G.Rodolico - San Marco, Catania
  - Fondazione Irccs Policlinico San Matteo, Pavia
  - EMATOLOGIA - Città della Scienza e Salute - Torino, Torino

IPD SHARING:
Plan to Share IPD: No